CLINICAL TRIAL: NCT06903104
Title: Acceptability and Feasibility of a Stress Prevention Program Based on Meditation and Acceptance and Commitment Therapy for Staff at a Cancer Center
Acronym: MAEva-pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02765-42
Record Dates: First submitted 2025-03-13; First posted 2025-03-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-03

CONDITIONS: Employees at a Hospital
Keywords: MAEva program; Quality of life; Mindfulness; Workplace; Caregivers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAEva program is delivered in a closed format (Experimental): MAEva program is delivered in a closed format. One session per week for 3 weeks.
  Interventions: Other: Mindfulness closed program; Diagnostic Test: Quality of life evaluation; Diagnostic Test: Perceived Stress Scale; Diagnostic Test: Multidimensional Psychological Flexibility Inventory; Other: satisfaction questionnaire and semi-structured interview

INTERVENTIONS:
Other: Mindfulness closed program — MAEva program will be proposed with meditative practices and three different themes will be addressed (one theme per session): Meditation, Acceptance and Commitment to values.
Diagnostic Test: Quality of life evaluation — The assessment will be carried out at inclusion and after completion of the program.
Diagnostic Test: Perceived Stress Scale — The assessment will be carried out at inclusion and after completion of the program.
Diagnostic Test: Multidimensional Psychological Flexibility Inventory — The assessment will be carried out at inclusion and after completion of the program.
Other: satisfaction questionnaire and semi-structured interview — The assessments will be carried out after completion of the program.

SUMMARY:
The MAEva program seems to meet the challenges of implementing meditation for cancer care workers. As part of our Quality of Life and Working Conditions initiative, the investigator decided to offer it to staff at our Cancer Center. The MAEva program is delivered in a closed format: participants commit to following, as far as possible, the three sessions of the program - one session per week for 3 weeks. During the sessions, it will be proposed to train meditative practices and three different themes will be addressed (one theme per session): Meditation, Acceptance and Commitment to values.

Before and after the program, participants will complete a quality of life evaluation, a perceived stress scale, and a questionnaire to assess psychological flexibility.

At the end of the program, each participant will be asked to complete a satisfaction questionnaire and a semi-directive interview, by videoconference, or by telephone in the event of digital impossibility with voice recording, to enable a qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant of legal age
* Willingness to participate in the program - voluntary registration
* Commitment to attend all 3 program sessions
* Schedule compatible with participation in the 3 program sessions
* Participant has understood, signed and dated the consent form
* Participant affiliated to the social security system

Exclusion Criteria:

* No desire to participate in the program - non-registration
* Previous participation in MAEva program
* No commitment to participate in the 3 program sessions
* Agenda incompatible with the 3 program sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility and acceptability of the MAEva program among employees at a hospital (CLCC: Centre de Lutte Contre le Cancer or Cancer Center). | 5 weeks
  Participation rate of employees at a hospital in the MAEva program and number of sessions attended (number of participants who completed the entire program)
Evaluate the feasibility and acceptability of the MAEva program among employees at a hospital (CLCC: Centre de Lutte Contre le Cancer or Cancer Center). | 5 weeks
  Number of sessions attended (number of participants who completed the entire program)

SECONDARY OUTCOMES:
Evaluate the initial effectiveness of the MAEva program on the well-being of employees at a hospital. | 5 weeks
  Quality of working life assessment (subjective score between 1 and 10 on the Quality of Working Life Scale)
Evaluate the initial effectiveness of the MAEva program on the well-being of employees at a hospital. | 5 weeks
  Stress assessment (Perceived Stress Scale - PSS-10)
Evaluate the initial effectiveness of the MAEva program on the well-being of employees at a hospital. | 5 weeks
  Assessment of psychological flexibility (Multidimensional Inventory of Psychological Flexibility (MPFI-24))
Evaluate the initial effectiveness of the MAEva program on the well-being of employees at a hospital. | 5 weeks
  Assessment of participant satisfaction (subjective score between 1 and 10; open-ended questions (qualitative analysis))
Evaluate the initial effectiveness of the MAEva program on the well-being of employees at a hospital. | 5 weeks
  Assessment of processes at play during the intervention (semi-structured interviews (qualitative analysis))

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France